CLINICAL TRIAL: NCT05318417
Title: A Post-approval, Prospective, Nonrandomized, Single-arm Multicenter Investigation to Evaluate the Safety and Effectiveness of Cochlear Implantation in Children and Adults With Unilateral Hearing Loss/Single-sided Deafness
Brief Title: Investigation to Evaluate the Safety and Effectiveness of Cochlear Implantation in Children and Adults With Unilateral Hearing Loss/Single-sided Deafness
Acronym: PAS-SSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5816
Record Dates: First submitted 2022-03-17; First posted 2022-04-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss, Unilateral; Deafness, Unilateral
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Children and adults with unilateral hearing loss/single-sided deafness (Other)
  Interventions: Device: The Cochlear™ Nucleus® Cochlear Implant (CI) System

INTERVENTIONS:
Device: The Cochlear™ Nucleus® Cochlear Implant (CI) System — The Cochlear™ Nucleus® CI systems are designed to provide useful hearing. The system works by converting sound in the environment into electric pulses that stimulate the auditory nerve, allowing the brain to perceive sound. The Cochlear™ Nucleus® CI system has implanted and external components.
  Implanted component:
  The CI is surgically implanted under the skin behind the ear. It includes a receiver/stimulator to receive and decode the electrical signals from the sound processor and an electrode to deliver these signals to the cochlear.
  External components:
  The external components include a sound processor, and associated accessories and cables. The system is programmed by a Cochlear proprietary programming system, Custom Sound®.

SUMMARY:
The aim of the study is to assess the continued efficacy and safety of cochlear implantation in participants aged 5 years and above with Unilateral Hearing Loss (UHL)/Single Sided Deafness (SSD) supporting a change indication for use.

ELIGIBILITY:
Inclusion Criteria:

• Individuals 18 years or older (Group A)

Ear to be Implanted:

Severe sensorineural hearing loss (HL) defined as: Pure-tone average at 0.5, 1, 2, 4 kHz >80 dB HL ; Aided Consonant-Nucleus-Consonant Test (CNC) score ≤5% and

Normal Hearing Ear:

Normal or near normal hearing defined as an average of (0.5, 1, 2, 4kHz) ≤ 30 dB HL

• Children 5 years to 17 years, 11 months (Group B)

Ear to be Implanted:

Severe sensorineural HL defined as: Pure-tone average at 0.5, 1, 2, 4 kHz >80 dB HL; Aided CNC score ≤5% and

Normal Hearing Ear:

Normal or near normal hearing defined as an average of (0.5, 1, 2, 4kHz) ≤ 30 dB HL

* Previous experience with a current conventional treatment option for unilateral [SSD] HL (HA, bone-conduction device, or CROS technology), if no previous experience a minimum trial period of two weeks is required
* English spoken as a primary language
* Willing and able to provide written informed consent

Exclusion Criteria:

* Ossification, abnormal cochlear nerve or any other cochlear anomaly that might prevent complete insertion of the electrode array
* Previous cochlear implantation
* Hearing loss of neural or central origin, including auditory neuropathy
* Duration of profound sensorineural HL >10 years per self-report
* Active / chronic middle-ear infection; conductive HL in either ear
* Medical or psychological conditions that contraindicate undergoing surgery as determined by the Investigator
* Unrealistic expectations on the part of the participant/family, regarding the possible benefits, risks, and limitations that are inherent as determined by the Investigator
* Evidence of and/or suspected cognitive or developmental concern
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child or sibling
* Cochlear employees or employees of Contract Research Organizations (CROs) or contractors engaged by Cochlear for the purposes of this investigation
* Pregnant or breastfeeding women
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in sentence in noise scores at 12 months post-activation in the binaural (CI and normal hearing (NH)) listening condition compared to preoperatively in the best listening (NH alone or NH and hearing aid) condition in 3 speaker configurations. | pre-implantation, 12 months post-activation
  Measured with the Bamford-Kowal-Bench Sentence in Noise test (BKB-SIN). List of sentences are presented at 65 dBA with the level of noise varied stepwise at fixed signal to noise ratio to obtain a Speech Reception Threshold (SRT) where participants are able to repeat key words 50% of the time. Score range is not specified as metric is adaptive; lower scores indicate better performance. The 3 speaker configurations are: speech front/noise front; speech front/noise to NH ear; speech front/noise to poorer ear.
Number of procedure and device related adverse events classified by type, frequency and severity. | 36 months post-activation

SECONDARY OUTCOMES:
Change in participant reported spatial hearing at 12 months post-activation compared to pre-operative ratings. | pre-implantation, 12 months post-activation
  Assessed via Speech, Spatial, and Qualities of Hearing Scale (SSQ) questionnaire (parent or participant version dependent on age). Rating ranges from 0 (no ability) to 10 (complete ability). Higher scores indicate greater perceived abilities.
Change in word recognition at 12 months post-activation in the CI alone condition compared to preoperative aided condition in the poorer hearing ear alone. | pre-implantation, 12 months post-activation
  Measured via the Consonant-Nucleus-Consonant (CNC) Word Recognition Test. The score is the total number of words correct expressed as percent correct (range of 0-100); higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Crosson, Study Director — Cochlear
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Iowa, Iowa City, Iowa
  - New York Eye and Ear Infirmary, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Texas Southwestern Medical Center- Department of Otolaryngology Head and Neck Surgery, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.